CLINICAL TRIAL: NCT06302543
Title: Treatment of Premature Ovarian Insufficiency Using Autologous Bone Marrow Concentrates Through Transvaginal Approach Under Ultrasound Guidance
Brief Title: Treatment of Premature Ovarian Insufficiency Using Bone Marrow Cells
Acronym: alfarah
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: abdulmajeed hammadi (Industry)
Responsible Party: Sponsor-Investigator, abdulmajeed hammadi, clinical professor, Global Stem Cell Center, Baghdad
Organization: Global Stem Cell Center, Baghdad (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POI bone marrow
Record Dates: First submitted 2024-02-24; First posted 2024-03-08 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Premature Ovarian Insufficiency
Keywords: premature ovarian failure,bone marrow,treatment
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Intervention Model Description: single armed interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bone marrow (Experimental): autologous bone marrow derived mononuclear cells injected 1cc per ovary for 2 ovaries under general anesthesia under ultrasound guide
  Interventions: Procedure: autologous bone marrow cells injection

INTERVENTIONS:
Procedure: autologous bone marrow cells injection — under general anesthesia bone marrow aspiration done followed by cell concentration and transvaginal ovarian injection

SUMMARY:
investigator is doing single armed clinical interventional study to treat premature ovarian insufficiency with autologous bone marrow derived mononuclear cells to be given systematically and locally to the ovaries under ultrasound guidance with experienced gynecologist and to look for the results including: laboratory evidence through hormonal study ultrasound proof of ovarian follicle development. premature ovarian insufficiency is characterized by early loss of ovarian function (less than 40 years of age) manifested by menstrual irregularity or amenorrhea with elevated levels of gonadotropin hormones and low estrogen and anti-Mullerian hormone.

Autologous use of stem cells from bone marrow are alternative safe minimal manipulative products that can provide a solution to this clinical problem without the need for oocyte donation program.

DETAILED DESCRIPTION:
Premature ovarian insufficiency is a clinical syndrome characterized by early loss of ovarian function (less than 40 years of age) manifested by menstrual irregularity or amenorrhea with elevated levels of gonadotrophin hormones and low estrogen and anti-Mullerian hormone. The average age for menopause is 50-52 years in the developed world ,it is believed that about 1% for women less than 40 years of age and 0.1 in less than 30 years of age has premature ovarian insufficiency.

Etiology of POI may be genetic, chromosomal, or auto immune.in addition to cancer treatment and surgical causes.

Hormonal replacement therapy is recommended for POI patients to alleviate vasomotor symptoms in addition to prevent osteoporosis and ischemic heart disease.

Regenerative medicine is a new medical approach to treat variety of diseases involving many tissues or organs in human body using cells, biological products instead of drugs or physical factors.

Autologous use of stem cells from bone marrow or adipose tissue (stromal vascular fraction) or platelet rich plasma are alternative safe minimal manipulative products that can provide a solution to this clinical syndrome.

Only few cases had been mentioned in the literature offering autologous stem cells for treating POI including bone marrow or adipose derived stem cells in addition to mesenchymal stem cells expanded invitro.

the investigator use autologous bone marrow concentrate with transvaginal approach under ultrasound guidance to treat POI.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of premature Ovarian insufficiency.
2. ineffective hormonal therapy.
3. biochemical evidence of high gonadotropins.

Exclusion criteria:

1. solid or hematological malignancies.
2. bleeding disorders.
3. rejection of the procedure.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — mainly related to females
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
change in gonadotropin levels | check every 4 weeks through study completion, an average of 1 year".
  luteinizing hormone and follicular stimulating hormone are followed

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No